CLINICAL TRIAL: NCT04980898
Title: Randomized, Third-blind, Controlled Trial of Superiority (Versus Sequential Dressings Recommended by the HAS) of an Electrode Dressing (WoundEL® Electrostimulation Device) on the Healing of Venous Ulcers
Brief Title: Electrostimulation System WoundEL for Leg Ulcers Healing (
Acronym: ELEXICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature termination due to recruitment difficulties
Sponsor: CEN Biotech (Industry)
Collaborators: WoundEL Health Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1633
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Leg Ulcer; Electrical Remodeling
Keywords: WoundEL
MeSH Terms: conditions — Leg Ulcer; Atrial Remodeling

STUDY DESIGN:
Intervention Model Description: Superiority randomized controlled study, open label with blinded primary outcome assessor, multicentric
Who Masked: Outcomes Assessor
Masking Description: The third blind person will have photographs of the wound at 10 weeks and all the surface readings on tracing paper necessary for the automated calculation of the surface with specific software. Readings will be sent in random order and third parties will not know the treatment, patient or date of the reading.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electrical stimulation wound management system (Experimental): Two daily electrostimulation sessions using the WoundEL® device on wound two for 30 minutes at an adjustable intensity, between 5 and 42 milliampere and chosen by the patient.
  Interventions: Device: WoundEL medical device; Other: Standard cares
- Standard of care (Active Comparator): Use of dressings appropriate to the stage of healing according to French recommendations for the management of leg ulcers.
  Interventions: Other: Standard cares

INTERVENTIONS:
Device: WoundEL medical device — The WoundEl system is composed by: a class IIa device , a class IIb dressing electrode and a class I disperser electrode.
  Applied to the leg ulcer, WoundEL® reproduces the endogenous electrical current to stimulate all the factors contributing to healing. Electrical current is evenly spread over the Dressing Electrode which also maintains a moist wound healing environment.
  Arms: Electrical stimulation wound management system
Other: Standard cares — Cleaning and monitoring

SUMMARY:
Several studies have suggested that the endogenous electric field and its polarity stimulate the proliferation and migration of epithelial cells and therefore promote wound healing. WoundEL® will reproduce the endogenous electrical current to stimulate all the factors contributing to healing.

Electrostimulation of wounds, including the WoundEL® device, is a therapy listed but not yet reimbursed in France. The aim of this study is to show that the WoundEL® electrostimulation device is superior to the reference treatments recognized by the HAS.

DETAILED DESCRIPTION:
Patients with a leg ulcer will be randomized to the "usual treatment" or "WoundEL" group.

The progress of the leg ulcer will be monitored every 2 weeks for 8 weeks or sooner if wound healing occurs. All leg ulcers will be examined at 10 weeks to check for healing or the condition of the leg ulcer if it has not healed. A third-blind party will also assess the ulcer condition at 10 weeks, based on standardized photographs.

The consumption of analgesics, pain and quality of life will be compared in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Venous leg ulcer evolving for at least 3 months, the area of which is between 4 cm² and 200 cm² and the smallest axis of which is less than 10 cm and the largest axis less than 20 cm;
* Have a Systolic Pressure Index (IPS) at the ankle between 0.89 and 1.3 and / or a systolic pressure measurement at the big toe greater than or equal to 60 mmHg;
* Accept the port of venous compression;
* Presenting superficial and / or deep venous insufficiency, documented on a Doppler echo dating less than one year;
* affiliated to a social security scheme or beneficiary of such a scheme;
* Having given their free, informed and written consent.

Exclusion Criteria:

* Untreated infected wound;
* Cancerous ulcer;
* Treated with systemic corticosteroids or chemotherapy;
* for which a skin graft is necessary;
* Contraindications for the treatment of leg ulcers with the WoundEL system;
* Pregnant or lactating women;
* Vulnerable people or under legal/judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Rate of healed-leg ulcers | At week 8
  Complete wound-healing correspond to 100% epithelialization of the leg ulcer, without persistent erosion or crusting. Complete healing of ulcers will be observed by the investigator and assessed by a third-blind.

SECONDARY OUTCOMES:
Assessing the leg ulcer-related pain | At weeks 0,2, 4, 6, 8
  Visual Analogic Scale
Assessing the analgesic consumption | At weeks 0,2, 4, 6, 8
  Patient reported-consumption of painkillers
Assessing the quality of life | At weeks 0,2, 4, 6, 8
  EuroQol (EQ5-D) questionnaire
Assessing the leg ulcer healing stage | At weeks 0,2, 4, 6, 8, 10
  Area measurement, periwound skin aspect, local signs of infection, antibiotic rescue
WoundEL system security | At weeks 0,2, 4, 6, 8
  Adverse reactions, dysfunctions

CONTACTS AND LOCATIONS:
Overall Officials: HERVE MAILLARD, MD, Principal Investigator — Centre Hospitalier du Mans; LAURE-CECILE MARTIN, Study Director — WoundEL Health Care
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No